CLINICAL TRIAL: NCT06349850
Title: Predictive Value of Serum Uric Acid to High Density Lipoprotein Cholesterol Ratio for Diabetic Kidney Injury in Type 2 Diabetes
Brief Title: Predictive Value of Serum Uric Acid to HDL Cholesterol Ratio for Diabetic Kidney Injury in Type 2 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eldeeb Elsayed Mohamed, Eldeeb Elsayed Mohamed, Sohag University
Other Study IDs: Soh-Med-24-03-06MS
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Kidney Injury
Keywords: DKI

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HbA1c level group: * well controlled diabetic group : HBA1c less than 7%
  * poorly controlled diabetic group : HBA1c equal to ore more than 7%
  Interventions: Diagnostic Test: serum uric acid level to plasma HDL-c level ratio (UHR)
- UHR level group: median levels of UHR will be used to dichotomize the patients into groups of :
  * low UHR group
  * high UHR group
  Interventions: Diagnostic Test: serum uric acid level to plasma HDL-c level ratio (UHR)
- DKI group: study population will be grouped into another two groups according to the presence of DKI:
  * patients with DKI
  * patients without DKI
  Interventions: Diagnostic Test: serum uric acid level to plasma HDL-c level ratio (UHR)

INTERVENTIONS:
Diagnostic Test: serum uric acid level to plasma HDL-c level ratio (UHR) — high UHR is considered to be a risk factor for development of DKI in type 2 DM

SUMMARY:
An prospective observetional study to asses the predictive value of serum uric acid to high density lipoprotein cholesterol ratio for diabetic kidney injury in type 2 diabetes

DETAILED DESCRIPTION:
Diabetic Kidney Injury (DKI) is a serious microvascular complication of diabetes mellitus occuring in about 20 % to 50% of diabetic patients and is the single commonest cause of ESRD.DKI is asociated with arterial HTN and increased cardiovascular morbidity and mortality. outcomes for both type 1 DM and type 2 DM who develop DKI are significantly worse than who do not .Serum uric acid was reported to be asociated with inflamatory and metabolic diseases such as metabolic syndrome , type 2 DM,thyroiditis and NAFLD while HDL-cholesterol decreased the odds of developing DKI by 20%.It is generally accepted that hyperuricemia and low HDL-c were considered to be a risk factor of other indicators for development of DKI.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* willing and agreed to be included in the study

Exclusion Criteria:

* Type 1 DM patients
* patients with active urinary sediment
* patients with glomerulonephritis
* patients with diagnosis or clinical features that are suspicious for another systemic disease that commonly causes kidney disease
* patients with evidence of alternative kidney disease
* patients with history of kidney transplantation
* patients with end stage renal disease
* patients with family history of non diabetic forms of kidney disease
* patients with active malignancy
* patients with established hemolytic disease
* CKD patients requiring dialysis
* patients taking drugs that interfere with serum uric acid level
* patients taking drugs that alter serum lipids level
* pregnancy
* Refused to consent to this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we will prospectively enroll patients from internal medicine department from march 2024 to august 2024 .all patients will be subjected to
  1. Detailed medical history including : demographic characteristics,comorbid conditions,duration of diabetes mellitus,type of treatment and diabetic complications
  2. Detailed clinical examination including : height , weight ,waist circumferenc,SBP,DBP,BMI
  3. Fundus examination for retinopathy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Uric acid to HDL-c ratio (UHR) | 6 months
  asociation of high UHR with development of DKI in type 2 DM

CONTACTS AND LOCATIONS:
Overall Officials: Eldeeb E. Mohamed, Principal Investigator — Sohag University

REFERENCES:
- [Background] Evans K, Pyart R, Steenkamp R, Whitlock T, Stannard C, Gair R, McCann J, Slevin J, Medcalf J, Caskey F. UK Renal Registry 20th Annual Report: Introduction. Nephron. 2018;139 Suppl 1:1-12. doi: 10.1159/000490958. Epub 2018 Jul 10. No abstract available. PMID 29990996
- [Background] Koye DN, Shaw JE, Reid CM, Atkins RC, Reutens AT, Magliano DJ. Incidence of chronic kidney disease among people with diabetes: a systematic review of observational studies. Diabet Med. 2017 Jul;34(7):887-901. doi: 10.1111/dme.13324. Epub 2017 Mar 9. PMID 28164387
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Diabetes and CKD: 2012 Update. Am J Kidney Dis. 2012 Nov;60(5):850-86. doi: 10.1053/j.ajkd.2012.07.005. PMID 23067652